CLINICAL TRIAL: NCT00079625
Title: Allogeneic Breast Protocol 2: Phase I Trial of T Cell Exchange With Th2/Tc2 Cells for Allogeneic Stem Cell Transplantation After Reduced Intensity Conditioning for Metastatic Breast Cancer
Brief Title: Stem Cell Transplant With Th2/Tc2 Cells to Treat Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040131; 04-C-0131; NCT00082953 (obsolete NCT alias)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-08-09

CONDITIONS: Breast Neoplasms
Keywords: Engraftment; Graft-Versus-Host Disease; Metastatic Breast Cancer; MBC
MeSH Terms: conditions — Breast Neoplasms; Graft vs Host Disease

INTERVENTIONS:
Drug: Th2/Tc2 Cells

SUMMARY:
This Phase 1 trial will investigate the safety of a modified stem cell transplant procedure for treating advanced breast cancer. Patients with cancers can sometimes benefit greatly from transplants of stem cells (cells produced by the bone marrow that mature into blood cells). In addition to producing new bone marrow and restoring normal blood production and immunity, the donated cells fight any residual tumor cells that might have remained in the body, in what is called a "graft-versus-tumor" effect. However, severe problems, or sometimes even death, may follow these transplants as a result of the high-dose chemotherapy and radiation that accompany the procedure. Also, donated immune cells called lymphocytes, or T cells, sometimes attack healthy tissues in a reaction called graft-versus-host-disease (GVHD), damaging organs such as the liver, intestines and skin. This study will use the following strategies to try to reduce these risks:

* "Induction chemotherapy" to reduce patients' immunity in an attempt to prevent rejection of the donated stem cells
* Reduced-intensity conditioning chemotherapy that is easier for the body to tolerate and involves a shorter period of complete immune suppression
* Removal of lymphocytes from the donor stem cells for transfusion in small quantities at monthly intervals following the stem cell transplant to reduce the risk of GVHD
* Transplant of specific lymphocytes called Th2/Tc2 cells that may increase the percentage of donor stem cells accepted by the patient without significantly increasing GVHD

Patients between 18 and 75 years of age with advanced (stage IV) breast cancer that does not respond to standard therapy may be eligible for this study. Candidates are screened with a medical history, physical and dental examinations, x-ray studies and bone marrow biopsies to evaluate disease status, blood and urine tests (including a blood test for genetic match with the donor), and lung and heart function tests.

Participants have a central venous line (large plastic tube) placed into a major vein. This tube stays in the body during the entire treatment period for infusing the donated stem cells and T lymphocytes, giving medications, including chemotherapy and other drugs, antibiotics, and blood transfusions, and withdrawing blood samples. Treatment starts with induction chemotherapy, in which patients receive one or two cycles of the anti-cancer drugs fludarabine and cyclophosphamide. (One cycle consists of 4 days on drug therapy followed by a 17-day rest period.) G-CSF, a drug that boosts white cell production, is also given to reduce the risk of infection. Several days before the transplant procedure, patients begin conditioning chemotherapy with higher doses of cyclophosphamide and fludarabine. Three days after the conditioning therapy is completed, the stem cells are infused. To help prevent both rejection of the donor stem cells and GVHD, patients receive cyclosporine (first by vein and later by mouth) for several weeks after the transplant. Infusions of donor lymphocytes begin about 6 weeks after the transplant to boost the immune system and enhance the graft-versus-tumor effect.

Patients may leave the hospital when they are able to eat and drink, have no fever or infection, and have a normal or near-normal white cell count. They return for follow-up visits twice a week for the first 100 days after the transplant, then every 3 months, then 6 months and then yearly for at least 5 years post-transplant. The visits include a medical history, physical examination, and blood draws, as well as disease staging with CT scans every month for the first 6 months.

DETAILED DESCRIPTION:
Background:

* In CC# 00-C-0119 we were able to demonstrate that allogeneic T cells could mediate a clinically relevant graft-versus-tumor (GVT) effect against MBC after a reduced-intensity, T cell depleted allogeneic hematopoietic stem cell transplant (alloHSCT).
* Responses were observed after establishment of complete lymphoid chimerism, which was frequently delayed and required the use of planned donor lymphocyte infusions (DLI). DLI were associated with a significant incidence of graft-versus-host disease (GVHD).
* In murine models, in vitro generated T cells of Th2/Tc2 phenotype can facilitate engraftment of HLA disparate allografts with significantly reduced GVHD as compared to T cell replete allografts that have not been manipulated. In addition, Th2/Tc2 cells provide an anti-tumor effect through the perforin/granzyme pathway.
* Allogeneic Th2/Tc2 cells may facilitate rapid allo-engraftment post-transplant with reduced GVHD. In addition, the perforin-mediated anti-tumor activity of Th2/Tc2 cells should provide earlier benefit compared with T-cell depleted allografts.

Objectives:

-To determine the safety, as defined by the incidence of acute graft-versus-host disease, and feasibility of administering in vitro generated donor T cells of Th2/Tc2 phenotype to augment a T cell depleted allograft (T cell exchange) after reduced-intensity conditioning.

Eligibility:

* Patients with measurable, metastatic breast cancer and an HLA matched sibling donor
* Patients must have received treatment with a taxane, an anthracycline, a hormonal agent and/or Herceptin, if the tumor expresses the respective receptors, and at least one treatment for metastatic disease that has not resulted in a complete response.

Design:

* Donors will initially have lymphocytes collected to generate the Th2/Tc2 product and then have blood stem cells collected following mobilization with filgrastim. The stem cell product will be T-cell depleted, and the T-cell dose will be adjusted to 1 x 10(5) CD3+ cells/kg.
* Patients will receive induction (immune depleting) chemotherapy with the goal of reducing circulating CD4+ cell less than 50/microliter prior to proceeding to alloHSCT.
* Patients will receive a reduced-intensity conditioning regimen consisting of fludarabine and cyclophosphamide. This will be followed by infusion of the T cell depleted allograft, which will be supplemented with Th2/Tc2 cells (i.e. T cell exchange).
* Cyclosporine will be discontinued after 40 days to permit a full GVT effect. Patients may receive donor lymphocyte infusions at days +42, +70, +98 post-transplant to further potentiate a GVT effect.
* Patients will be enrolled in three cohorts, with escalating Th2/Tc2 cell doses (0.5 - 12.5 x 10(7) cells/kg) given in a phase-I manner.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria - Recipient:

1. Patients with measurable stage IV breast cancer. Patients with central nervous system CNS metastases are eligible if the CNS metastases have been treated and remained stable a minimum of four weeks after the completion of therapy.
2. Patients must have received at least one prior chemotherapy regimen for treatment of distant metastases and achieved less than a complete response to this therapy.

   1. Patients must have received prior therapy with a taxane (e.g. paclitaxel) and an anthracycline (e.g. doxorubicin) as part of either adjuvant therapy or treatment of metastatic disease.
   2. Patients whose tumor expresses estrogen and/or progesterone receptors must have received at least one hormonal therapy (e.g. Tamoxifen) as part of either adjuvant therapy or treatment of metastatic disease.
   3. Patients whose tumor expresses Her2-neu must have received trastuzumab (Herceptin ) as part of either adjuvant therapy or treatment of metastatic disease.
   4. Patients who have undergone prior autologous stem cell transplantation are eligible for this protocol.
3. Patients 18 - 75 years of age. The upper age limit was chosen in order not to be discriminatory, provided that patients meet all other eligibility criteria.
4. ECOG performance status less than or equal to 2 (Karnofsky performance status greater than or equal to 60%).
5. Life expectancy greater than 6 months.
6. Left ventricular ejection fraction has to be greater than or equal to 45% by either MUGA or 2-D echo. This test will repeated immediately after induction and prior to transplantation. Patients who do not have the minimally required function will be removed from trial.
7. DLCO greater than or equal to 50% of the expected value when corrected for Hb. This test will repeated immediately after induction and prior to transplantation. Patients who do not have the minimally required function will be removed from trial.
8. Creatinine less than or equal to 1.5 mg/dl and a creatinine clearance greater than or equal to 50 ml/min/1.73 m(2). This test will repeated immediately after induction and prior to transplantation. Patients who do not have the minimally required function will be removed from trial.
9. Direct bilirubin less than or equal to 2.5 mg/dl, SGOT less than 4x high normal value. Values above these levels may be accepted, at the discretion of the PI or study chairperson, if such elevations are thought to be due to liver involvement by malignancy. This test will repeated immediately after induction and prior to transplantation. Patients who do not have the minimally required function will be removed from trial.
10. Patients must be HIV-, HbsAg-, and Hepatitis C antibody negative. The high degree of immune suppression that will be used in this study may lead to the activation or progression of these viral illnesses.
11. Not pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of the chemotherapy, the subsequent transplant and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are unknown and may be harmful to the infant.
12. Consenting sibling matched at 6/6 HLA antigens.
13. Provision for a Durable Power of Attorney.
14. Ability to give informed consent.

Inclusion Criteria - Donor:

1. Age 18 - 75 years. As the potential for cerebrovascular and cardiac complications may potentially increase with age, 75 years has been chosen arbitrarily as the upper age limit. However, if it is determined after initial accrual of patients in this upper age range that this procedure is relatively safe, the age range may be extended.
2. No physical contraindications to stem cell donation (i.e. severe atherosclerosis, auto-immune disease, cerebrovascular accident, prior malignancy. Patients with severe atherosclerosis by history will receive a cardiology consult and be judged eligible on a case by case basis. The exclusion of patients with a prior malignancy will be evaluated on a case by case basis. If it is felt by the investigators that the risk of potential transfer of malignant cells is far outweighed by the potential benefit of the procedure the patient may be eligible to serve as a donor. Persons with a history of non-hematologic malignancy must have undergone potentially curative therapy for that malignancy and 1) have had no evidence of that disease for 5 years, and/or 2) be deemed at low risk for recurrence (less than or equal to 20% at 5 years). Such persons will be considered eligible for stem cell donation at the discretion of the principal investigator, who will evaluate the possible benefit to the potential transplant recipient and the risk of disease transmission in consultation with Department of Transfusion Medicine staff. Prospective donors with a history of non-hematologic malignancy who have received potentially curative therapy and are in remission, but whose estimated risk of recurrence is greater than 20% at 5 years, will be considered on an individual basis in consultation with the NCI IRB. Any prospective transplant recipient whose donor has a history of malignancy will be counseled about the theoretical risk of transmission of cancer from the donor to the recipient.
3. Donors must be HIV-negative, HbsAg, and Hepatitis C antibody negative. As donors are providing an allogeneic blood product there is the potential risk of transmitting these viral illnesses to the recipient.
4. Donor must not be pregnant or breastfeeding an infant. A donor who is lactating must substitute formula feeding for her infant during the period of cytokine administration. Filgrastim may be secreted in human milk, although its bioavailability from this source is not known. Limited clinical data suggest that short-term administration of filgrastim or sargramostim to neonates is not associated with adverse outcomes. Donors of childbearing potential must use an effective method of contraception during the time they are receiving cytokines. The effects of cytokine administration on a fetus are unknown and may be potentially harmful. The effects upon breast milk are also unknown and may potentially be harmful to the infant.
5. Ability to give informed consent.

EXCLUSION CRITERIA:

Exclusion Criteria - Patient

1. Active infection that is not responding to antimicrobial therapy.
2. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent (as determined by principal investigator).

Exclusion Criteria - Donor

1. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
2. History of hypertension that is not controlled by medication, stroke, or severe heart disease. Individuals with symptomatic angina will be considered to have severe heart disease and will not be eligible to be a donor.
3. Anemia (Hb less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000 per ml).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-03-05; Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety as defined by the incidence of acute graft-versus-host disease and feasibility of administering in vitro generated donor T cells of Th2/Tc2 phenotype to augment a T cell depleted allograft after reduced-intensity conditio...

SECONDARY OUTCOMES:
To determine if the transplantation of a T cell depleted allograft augmented with Th2/Tc2 ell can result in a state of rapid complete donor chimerism after reduced-intensity conditioning regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Fowler, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nemoto T, Natarajan N, Bedwani R, Vana J, Murphy GP. Breast cancer in the medial half. Results of 1978 National Survey of the American College of Surgeons. Cancer. 1983 Apr 15;51(8):1333-8. doi: 10.1002/1097-0142(19830415)51:83.0.co;2-t. PMID 6825053
- [Background] Smith RE, Brown AM, Mamounas EP, Anderson SJ, Lembersky BC, Atkins JH, Shibata HR, Baez L, DeFusco PA, Davila E, Tipping SJ, Bearden JD, Thirlwell MP. Randomized trial of 3-hour versus 24-hour infusion of high-dose paclitaxel in patients with metastatic or locally advanced breast cancer: National Surgical Adjuvant Breast and Bowel Project Protocol B-26. J Clin Oncol. 1999 Nov;17(11):3403-11. doi: 10.1200/JCO.1999.17.11.3403. PMID 10550134
- [Background] Hortobagyi GN. Recent progress in the clinical development of docetaxel (Taxotere). Semin Oncol. 1999 Jun;26(3 Suppl 9):32-6. PMID 10426457
- [Derived] Hardy NM, Mossoba ME, Steinberg SM, Fellowes V, Yan XY, Hakim FT, Babb RR, Avila D, Gea-Banacloche J, Sportes C, Levine BL, June CH, Khuu HM, Carpenter AE, Krumlauf MC, Dwyer AJ, Gress RE, Fowler DH, Bishop MR. Phase I trial of adoptive cell transfer with mixed-profile type-I/type-II allogeneic T cells for metastatic breast cancer. Clin Cancer Res. 2011 Nov 1;17(21):6878-87. doi: 10.1158/1078-0432.CCR-11-1579. Epub 2011 Sep 26. PMID 21948234